CLINICAL TRIAL: NCT02107365
Title: Pilot Study to Assess Efficacy and Safety of a Quadruple Therapy With Asunaprevir, Daclatasvir, Ribavirin and Pegylated Interferon Alpha-2a in HCV Genotype 4-infected Patients Non-responders to Pegylated Interferon-Ribavirin Regimen
Brief Title: Therapy With Asunaprevir, Daclatasvir, Ribavirin and Pegylated Interferon Alpha-2a in HCV Genotype 4-infected Patients Who Have Failed to a Previous Therapy With Peg-Interferon/Ribavirin (ANRS HC32 QUATTRO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS HC32 QUATTRO
Record Dates: First submitted 2014-03-31; First posted 2014-04-08 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Hepatitis C Virus Genotype 4 Infection
Keywords: Hepatitis C; HCV infection; HCV genotype 4; Non-responders HCV infected patients; Asunaprevir; Daclatasvir; Pegylated Interferon; Ribavirin
MeSH Terms: conditions — Hepatitis C | interventions — asunaprevir; daclatasvir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Asunaprevir, Daclatasvir, Ribavirin, Peg-Interferon alpha-2a (Experimental): Quadritherapy from Day 0 to Week 24
  Interventions: Drug: Asunaprevir; Drug: Daclatasvir; Drug: Ribavirin; Drug: Pegylated Interferon alpha-2a

INTERVENTIONS:
Drug: Asunaprevir — Asunaprevir 100 mg, 1 capsule twice a day from Day 0 to Week 24
Drug: Daclatasvir — Daclatasvir 60 mg, 1 tablet once a day from Day 0 to Week 24
Drug: Ribavirin — Ribavirin tablets or capsules 200 mg, weight-based daily dose ( <75 kg : 1000 mg ; ≥ 75 kg : 1200 mg), from Day 0 to Week 24
Drug: Pegylated Interferon alpha-2a — Pegylated Interferon alpha-2a, by subcutaneous injection 180µg / week, from Day 0 to Week 24

SUMMARY:
Success rates, after retreatment with Peg-Interferon/Ribavirin bitherapy, in patients infected with HCV (hepatitis C virus) genotype 4 and non-responders to a first standard treatment, are disappointing. The association of Asunaprevir and Daclatasvir in combination with the standard-of-care bitherapy has been shown to increase the efficacy of the treatment in non-responders genotype 1-infected patients.

Given the absence of current solutions and urgent therapeutic needs for HCV genotype 4-infected patients previously treated with pegylated Interferon/Ribavirin, this pilot study aims to evaluate the efficacy and safety of a quadritherapy associating Asunaprevir, Daclatasvir, pegylated Interferon alpha-2a and Ribavirin, in this very difficult to treat population.

60 subjects will be enrolled.

The primary endpoint will be the rate of sustained virological response (SVR), defined by an undetectable HCV RNA, at Week 36 (12 weeks after the end of a 24 weeks quadritherapy).

DETAILED DESCRIPTION:
The population studied presents the maximum of factors of non-response to the retreatment of hepatitis C: non-response to well followed prior treatment with pegylated Interferon and Ribavirin, infection with HCV genotype 4, and the presence of cirrhosis (in less than 50% of the included patients) that could diminish the chances of SVR to a standard bitherapy.

The likelihood of SVR with standard bitherapy in this study population is thus considered low, around 15%.

The principal objective of this multicentric, national, single-arm, open-labeled, non-randomized phase II pilot study in 60 patients, is to assess the rate of SVR 12 weeks after 24 weeks of quadritherapy and to determine whether this rate is significantly greater than 20%.

The proportion of patients presenting with cirrhosis (defined by a METAVIR F4 score on liver biopsy or with hepatic impulse elastometry ≥ 15 kPa) will be limited to 50% of all patients included.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years
* Infection with HCV genotype 4, confirmed by detectable HCV RNA ≥ 1000 IU/ml at pre-inclusion
* Non-responders to a prior treatment with pegylated Interferon and Ribavirin, with non-response being defined as follows:

  * Null-response: reduction of less than 2 log10 IU/ml of HCV viral load between D0 of the treatment and week 12
  * Partial response: reduction of at least 2 log10 IU/ml of HCV viral load between D0 of the treatment and week 12 but detectable HCV RNA at week 12 and week 24 and without an undetectable viral load by the end of treatment
* Anti-HCV treatment discontinued for at least the last 3 months
* Fibrosis at any stage, with documentation of the presence or absence of cirrhosis at the pre-inclusion visit:

  * history of liver biopsy showing cirrhosis lesions (METAVIR F4), at any time in the patient's history, and/or
  * good quality (length ≥ 15 mm and ≥ 6 portal spaces) liver puncture biopsy from less than 18 months to establish the METAVIR, and/or
  * hepatic impulse elastometry (Fibroscan®) from less than 6 months and of good quality (at least 10 measurements on an incidence with an IQR of less than 30% of the mean elastometry measured and a success rate of 60%)
* Body weight ≥ 40 kg and ≤125 kg
* Men and women of child-bearing age and their heterosexual partners must use two adequate contraceptions from 1 month before initiation of treatment up to 7 months after the end of treatment for men and up to 4 months after treatment for women.
* Written informed consents (2) signed by the patient and the investigator (on the day of the pre-inclusion at the latest and before any examination required by the study)
* Patients with Health insurance (Sécurité Sociale or Couverture Médicale Universelle)

Exclusion Criteria:

* CHILD B or C cirrhosis or a history of decompensated cirrhosis. If Child A cirrhosis, presence of varices presenting an hemorrhagic risk (grade II with red spots or grade III) on a fibroscopy dating from less than 3 years
* Previous HCV therapy including HCV NS3 protease inhibitor, and/or HCV NS5A replication complex inhibitor and/or HCV NS5B polymerase inhibitor
* Positive HBs Antigen
* Confirmed HIV-1 or HIV-2 infection
* Pregnant or breast-feeding women
* Severe heart or lung disease
* Transplant recipient
* Uncontrolled dysthyroidism
* Uncontrolled diabetes
* Any evolutive ongoing malignant disease, including hepatocellular carcinoma, which will be specifically screened for before inclusion
* Consumption of alcohol which, in the opinion of the investigator, will be an obstacle to participation of the patient and to his remaining in the study
* Drug addiction which, in the the investigator's opinion, will be an obstacle to the patient's participation and to his or her remaining in the study. Patients included in a programme of substitution with methadone or buprenorphine could be included. The opinion of a consultant in addictology is recommended for patients presenting with current drug use or drug use in the past year.
* Patients taking part in another clinical trial during the 30 days preceding inclusion.
* Patient under guardianship, trusteeship or judicial protection
* Hb < 110 g/L
* Platelets < 80 000/mm3
* Polynuclear neutrophils < 1000 /mm3 (for European patients) and < 750 /mm3 (for African patients)
* Kidney failure defined by creatinine clearance < 50mL/mn (MDRD formula)
* Contra-indication for treatment with Ribavirin including a history of hypersensitivity to Ribavirin or to one of the excipients
* Contra-indication for treatment with Daclatasvir or Asunaprevir including a history of hypersensitivity to one of the excipients
* Contra-indication to treatment with Interferon including psychiatric contra-indications. A psychiatrist's opinion is compulsory in the following situations :

  * history of psychiatric disorders requiring hospitalisation of the patient or a consultation with a specialist
  * treatment with mood stabilizers or antipsychotics during the previous year
  * history of psychiatric disorders during prior treatment with Interferon alpha
  * evidence of depression episodes, a risk of suicide, bipolar disorder and/or current behavioral disorders. These patients can only be included after a psychiatric evaluation that specifically authorizes the use of Interferon.
* History of previous HCV treatment premature cessation (in the first 6 months) for toxicity. Premature cessation for anemia or neutropenia will be authorized in the absence of the use of erythropoietin or polynuclear neutrophil growth factor, respectively.
* Patients with a non-compliance history, who will be at risk of not complying with the study follow-up timetable
* Associated treatment likely to interfere with the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
SVR12 Rate | Week 36
  HCV RNA measured 12 weeks after the end of the HCV treatment (Week 36)

SECONDARY OUTCOMES:
Number of patients with adverse events | Up to Week 48
Treatment discontinuations | Up to Week 24
  Number and causes of treatment discontinuations
Self-reported symptoms | Day 0, Week 12, Week 36
  ANRS AC24 perceived symptoms scale
Patients' adherence | Week 4, Week 12, Week 24
  ANRS questionnaire
SVR 24 rate | Week 48
  Undetectable HCV RNA 24 weeks after the end of the HCV treatment
HCV viral load | Day 0, Weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 36, 48
Number of patients with virological failure under treatment | Up to Week 24
  Patients with detectable HCV viral load at Week 8, or Patients with HCV breakthrough : a) undetectable HCV viral load at Week 8 and detectable at any visit after Week 8 or b) undetectable HCV viral load at any time point before Week 8 and who presents a new confirmed detectable viral load before Week 8
HCV subtypic distribution | Baseline
Proportion of patients with resistance mutations to Asunaprevir and/or Daclatasvir in case of virological failure | Up to Week 48
Cirrhosis evaluation | Baseline, Week 12, Week 24, Week 36, Week 48
  For cirrhotic patients : Child-Pugh and MELD scores ; cirrhosis decompensation evaluation on clinical examination
Insulin resistance : HOMA-IR score | Day 0, Week 36
Metabolic syndrome parameters | Day 0, Week 36
  Waist circumference, blood pressure, fasting glucose, triglycerides, HDL cholesterol (composite measure)
Liver fibrosis | Between baseline and Week 48
  Evolution of liver fibrosis on biological parameters (Fibrotest®) and imaging (Fibroscan®)
Polymorphism of the gene of IL28B | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Dominique ROULOT, MD, PhD, Principal Investigator — Bobigny University Hospital; Eric BELLISSANT, MD, PhD, Study Chair — Rennes University Hospital
Locations (25):
- France (25):
  - Hôpital AVICENNE, Bobigny
  - Hôpital Jean Verdier, Bondy
  - Hôpital de Haut Lévêque, Bordeaux Pessac
  - Hôpital Beaujon, Clichy
  - Centre Hospitalier Intercommunal, Créteil
  - Hôpital Henri Mondor, Créteil
  - Hôpital Albert Michallon, Grenoble
  - Hôpital Claude Huriez, Lille
  - Hôpital Dupuytren, Limoges
  - Hôpital de la Croix Rousse, Lyon
  - Fondation Hôpital Saint Joseph, Marseille
  - Hôpital Saint Eloi, Montpellier
  - Hôpital de Brabois, Nancy
  - Hôpital de l'Hôtel Dieu, Nantes
  - Hôpital de l'Archet, Nice
  - Hôpital de La Source, Orléans
  - Hôpital Saint Antoine, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Cochin, Paris
  - Hôpital Tenon, Paris
  - Hôpital Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Institut Arnault Tzank, Saint-Laurent-du-Var
  - Hôpital Purpan, Toulouse
  - Hôpital Paul Brousse, Villejuif